CLINICAL TRIAL: NCT06936618
Title: Using Electrical Impedance Tomography-Guided Ventilator Settings to Reduce Mechanical Power in Acute Hypoxemic Respiratory Failure : An Exploratory Study
Brief Title: EIT-Guided Ventilator Settings in AHRF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SI 962/2024
Record Dates: First submitted 2025-03-26; First posted 2025-04-20 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Hypoxemic Respiratory Failure; Acute Respiratory Distress Syndrome (ARDS); Mechanical Power; Ventilator Induced Lung Injury; Electrical Impedance Tomography (EIT)
Keywords: Acute Hypoxemic Respiratory Failure; Electrical Impedance Tomography; Mechanical Power, Ventilator-induced lung injury
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Ventilator-Induced Lung Injury

STUDY DESIGN:
Intervention Model Description: All enrolled patients will receive the intervention using EIT-guided PEEP titration. Outcomes such as mechanical power, lung mechanics, and gas exchange will be measured before and after the intervention in a single-arm, pre-post study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EIT-guided PEEP titration (Experimental): Patients will undergo ventilator adjustments using EIT-guided PEEP titration to optimize mechanical power and lung mechanics.
  Interventions: Device: Electrical Impedance Tomography (EIT), Enlight 2100

INTERVENTIONS:
Device: Electrical Impedance Tomography (EIT), Enlight 2100 — Patients will undergo ventilator adjustments using EIT-guided PEEP titration to optimize mechanical power and lung mechanics.

SUMMARY:
This exploratory study aims to investigate the effect of Electrical Impedance Tomography (EIT)-guided ventilator settings on mechanical power in patients with acute hypoxemic respiratory failure (AHRF), including both ARDS and non-ARDS conditions. Mechanical power, a key factor associated with ventilator-induced lung injury (VILI), will be measured before and after EIT-guided PEEP titration. The study will evaluate feasibility and changes in lung mechanics, gas exchange, and EIT parameters. A total of 17 patients requiring invasive mechanical ventilation will be enrolled at Siriraj Hospital, Mahidol University.

DETAILED DESCRIPTION:
This exploratory study investigates the effect of Electrical Impedance Tomography (EIT)-guided PEEP titration on mechanical power in patients with acute hypoxemic respiratory failure (AHRF), including both ARDS and non-ARDS conditions such as severe pneumonia and pulmonary edema. Mechanical power represents the energy transferred from the ventilator to the respiratory system per unit time and has been associated with the development of ventilator-induced lung injury (VILI).

Patients who meet the inclusion criteria will undergo a standardized EIT-guided PEEP titration protocol using the Enlight 2100 EIT device. Optimal PEEP is defined as the PEEP level that minimizes both alveolar overdistension and collapse based on real-time EIT measurements. Mechanical power and other ventilatory parameters (lung compliance, plateau pressure, driving pressure, 4∆P x RR index, and gas exchange) will be assessed before and after PEEP titration at predefined time points (baseline, 2, 12, and 24 hours).

The study also evaluates the regional ventilation distribution ratios, as well as safety outcomes including hemodynamic instability, arrhythmias, and pneumothorax. Patients will be followed for up to 28 days to record duration of mechanical ventilation, ICU stay, and 28-day mortality.

This study aims to assess the feasibility and physiological benefits of personalized ventilator settings using EIT in critically ill patients with AHRF and to generate preliminary data for future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with acute hypoxemic respiratory failure within 48 hours
* Expected to require invasive mechanical ventilation ≥ 48 hours
* On mechanical ventilation within 24 hours
* Deep sedation and neuromuscular blockade

Exclusion Criteria:

* Pregnancy
* Body mass index (BMI) > 40 kg/m2
* Contraindications to using electrical impedance tomography, including
* Presence of a pacemaker or automatic implantable cardioverter-defibrillator (AICD)
* Inability to place the belt due to presence of surgical wounds dressing, thoracic or spinal cord trauma, recent thoracic surgery, etc.
* High risk for PEEP titration
* Hemodynamic instability defined as mean arterial pressure < 65 mmHg despite optimization of fluid status and/or use of vasopressors
* Unstable cardiac arrhythmias
* Presence of lung bullae greater than 2 cm in diameter, identified on chest X-ray
* Presence of pneumothorax or pneumomediastinum
* Right-sided heart failure or severe pulmonary hypertension
* Neurologic conditions associated with a risk of intracranial hypertension
* Use of extracorporeal membrane oxygenation (ECMO)
* Severe chronic respiratory disease, defined as follows: requiring home oxygen therapy, or previous lung function showing (FEV1 less than 20 ml/kg PBW, or FEV1/FVC less than 50% predicted value), or chronic hypercapnia (PaCO2 greater than 45 mmHg) and/or chronic hypoxemia (PaO2 less than 55 mmHg) on FIO2 = 0.21, or radiographic x-ray evidence of any chronic over-inflation or chronic interstitial infiltration, or chronic restrictive, obstructive, neuromuscular, chest wall or pulmonary vascular disease resulting in severe exercise restriction (unable to climb stairs or perform household duties, secondary polycythemia, severe pulmonary hypertension with mean pulmonary arterial pressure greater than 40 mmHg)
* Decision to withhold life-sustaining treatment or palliative care.
* Moribund status with an expected survival of less than 24 hours.
* Refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Mechanical Power | ฺBaseline and 2 hours after EIT-guided ventilator adjustment and follow-up over 24 hours (baseline, 2 hours, 12 hours, and 24 hours after EIT-guided ventilator adjustment)
  Mechanical power (MP) will be calculated using Gattinoni's simplified formula. Simplified Gattinoni's formula: MP = 0.098 × respiratory rate × tidal volume × [peak inspiratory pressure - (plateau pressure - PEEP)/2] calculated mechanical power (measured in J/min) before and after using EIT-guided PEEP titration in patients with acute hypoxemic respiratory failure.
  Unit of Measure: Joules per minute (J/min)

SECONDARY OUTCOMES:
Change in PEEP level | At baseline and then 2 hours, 12 hours, 24 hours after EIT-guided PEEP titration
  Positive End-Expiratory Pressure (PEEP) level before and after EIT-guided ventilator adjustment.
  Unit of Measure: cmH₂O
Change in Respiratory Static Compliance | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  calculate static respiratory compliance (tidal volume/driving pressure) before and after EIT-guided PEEP titration Unit of Measure: mL/cmH₂O
Change in Driving Pressure | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  calculate driving pressure (plateau pressure - PEEP) following EIT-guided PEEP titration.
  Unit of Measure: cmH₂O
Change in Plateau Pressure | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  measure plateau pressure before and after EIT-guided PEEP titration.
Change in 4∆P + RR Index | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  Calculated value of 4 x Driving Pressure + Respiratory Rate before and after EIT-guided PEEP titration.
  Unit of Measure: Joules per minute (J/min)
Change in Elastic dynamic power | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  calculate elastic dynamic power formula : elastic dynamic power = 0.098 x respiratory rate x tidal volume x 0.5 x driving pressure before and following EIT-guided PEEP titration Unit of Measure: Joules per minute (J/min)
change in elastic static power | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  calculated value of elastic static power = 0.098 x respiratory rate x tidal volume x PEEP before and after EIT-guided PEEP titration Unit of Measure: Joules per minute (J/min)
Change in resistive power | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  calculated resistive power = 0.098 x respiratory rate x tidal volume x (peak inspiratory pressure - plateau pressure) before and after EIT-guided PEEP titration Unit of Measure: Joules per minute (J/min)
Change in arterial oxygen tension (PaO₂) | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  Arterial oxygen tension (PaO₂) measured by arterial blood gas analysis before and after EIT-guided PEEP titration.
  Unit of Measure: PaO₂: mmHg
Ventilation distribution ratio | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  record anterior/posterior and right/left ventilation distribution from EIT before and after EIT-guided PEEP titration Unit of Measure: Percentage (%)
Incidence of complication | Up to 24 hours after intervention
  Number of patients experiencing adverse events related to EIT or ventilator adjustments, including pneumothorax, hemodynamic instability, or arrhythmia.
  Unit of Measure: Number of participants with event
Change in arterial carbon dioxide tension (PaCO₂) | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  Carbon dioxide tension (PaCO₂) measured by arterial blood gas analysis before and after EIT-guided PEEP titration.
  Unit of Measure: PaCO₂: mmHg
Change in arterial pH | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  Arterial pH measured by arterial blood gas analysis before and after EIT-guided PEEP titration.
  Unit of Measure: pH: unitless
Change in PaO₂/FiO₂ ratio | Baseline, 2 hours, 12 hours, and 24 hours after intervention
  PaO₂/FiO₂ ratio changes before and after EIT-guided PEEP titration. PaO₂/FiO₂ ratio will be calculated using PaO₂ from arterial blood gas and FiO₂ obtained from ventilator settings.
  Unit of Measure: PaO₂/FiO₂: mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ranistha Ratanarat, Associated Professor, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data.